CLINICAL TRIAL: NCT03397173
Title: Targeting TET2 Mutations in Myelodysplastic Syndromes and Acute Myeloid Leukemia (AML) With Azacitidine and Ascorbic Acid
Brief Title: TET2 Mutations in Myelodysplastic Syndromes and Acute Myeloid Leukemia With Azacitidine + Ascorbic Acid
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE1917
Record Dates: First submitted 2018-01-05; First posted 2018-01-11 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-08

CONDITIONS: Myelodysplastic Syndromes; Myeloproliferative Neoplasm; Acute Myeloid Leukemia
Keywords: Azacitidine; Ascorbic Acid
MeSH Terms: conditions — Myelodysplastic Syndromes; Myeloproliferative Disorders; Leukemia, Myeloid, Acute | interventions — Azacitidine; Ascorbic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Azacitidine + Ascorbic acid (Experimental): Azacitidine will be administered intravenously or subcutaneously at a fixed dose of 75mg/m2/day for 7 consecutive days, (allowing for weekends, and holidays) of each 28-day cycle. Ascorbic acid will be administered orally daily at 1 g/day three days prior to start azacitidine and then continues daily for a total of 28 days of each 28 day cycle.
  Interventions: Drug: Azacitidine; Drug: Ascorbic acid

INTERVENTIONS:
Drug: Azacitidine — Azacitidine will be administered intravenously or subcutaneously at a fixed dose of 75mg/m2/day for 7 consecutive days, allowing interruptions for weekends and holidays within each 28-day cycle. No dose modifications will be permitted during the treatment period.
Drug: Ascorbic acid — Ascorbic acid will be administered orally daily at 1 g/day three days prior to start azacitidine and then continues daily for a total of 28 days of each 28 day cycle. No dose modifications will be permitted during the treatment period.

SUMMARY:
The purpose of this study is to evaluate the efficacy of treatment with azacitidine (an FDA approved drug for the treatment of MDS) and high dose ascorbic acid in patients with TET2 mutations. This approach is intended to enhance the enzymatic activity of TET2 protein, which in term may help to improve counts and symptoms, related to Myelodysplastic Syndromes and Acute Myeloid Leukemia. This combination is specific to individuals who carry this mutation.

DETAILED DESCRIPTION:
Primary Endpoint To estimate the overall response rate (ORR) of the combination of standard dose azacitidine and oral dose of ascorbic acid in patients with MDS, AML, and MDS / Myeloproliferative Neoplasm (MPN) overlap with heterozygous TET2 mutations

Secondary Endpoints

1. The safety profile of the combination in the targeted patient population
2. Response duration
3. Overall survival of the treated population (compared to matched historical cohort of patients treated with single agent Azacitidine)
4. The identification of biomarkers that predict response to the combination

Study Design This is an open-label, phase II study that will be conducted at Cleveland Clinic, Taussig Cancer Institute.

Azacitidine will be administered intravenously or subcutaneously at a fixed dose of 75mg/m2/day for 7 consecutive days, (allowing for weekends, and holidays) of each 28-day cycle. Ascorbic acid will be administered orally daily at 1 g/day three days prior to start azacitidine and then continues daily for a total of 28 days of each 28 day cycle.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a confirmed heterozygous TET2 mutations identified by next generation targeted deep sequencing.
* Patients must have MDS, or MDS/MPN overlap defined by 2016 World Health Organization (WHO) criteria. Both newly diagnosed or previously treated MDS or MDS/MPN patients are eligible as long as the patient has never received prior treatment with azacitidine or decitabine.
* Patients with Leukemic/blast phase transformation MPN.
* Patient with AML according to 2016 WHO criteria.

  * Newly diagnosed patients who are ineligible or declined to receive intensive chemotherapy after discussion of risks and benefits of that approach or patients with primary refractory/relapsed AML.
  * Patients with active central nervous system (CNS) leukemia eligible at the discretion of treating physician.
  * Relapse/Refractory is defined as at least 1 course of treatment for AML excluding any patients treated with azacitidine or decitabine.

    * Patients should be off any prior treatment or line of therapy for 2 weeks prior to start study with the exception of hydrea (Hydroxyurea).
* Prior therapy with hydroxyurea, biological or targeted therapy (e.g. flt3 inhibitors, other kinase inhibitors) or hematopoietic growth factors is allowed.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 3.
* Patients must have normal organ and marrow function as defined at the discretion of the treating physician and PI.
* Women of childbearing potential must have a negative serum or urine pregnancy test within 10-14 days prior to enrollment.
* Patients must have the ability to understand and the willingness to sign a written informed consent document.
* Patient must be willing to comply with all aspects of the protocol including completing the drug diary.
* Patient must discontinue any and all use of multivitamin and/or vitamin c medication 24 hours before first dose of Ascorbic Acid.

Exclusion Criteria:

* Any prior treatment with azacitidine or decitabine.
* Patients diagnosed with acute promyelocytic leukemia (APL), AML-M3.
* Patients receiving other active treatment for their myeloid malignancy including investigational agents with the exception of hydrea for white blood cell control.
* Nursing or pregnant women.
* History of allergic reactions to either azacitidine or ascorbic acid.
* Patients with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients with higher risk of bleeding (deemed by the treating physician) or on anticoagulation.
* Patients who are unwilling or unable to comply with all study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-03-16 (Actual); Primary Completion 2021-01-03 (Actual); Study Completion 2021-01-21 (Actual)

PRIMARY OUTCOMES:
Number of patients with response per MDS International Working Group 2006 Criteria | 171 Days (6 cycles of 28 days plus 3 day loading period)
  A binary indicator of overall response, defined as achieving CR, PR, or HI) per 2006 International Working Group (IWG) criteria
  Responses for MDS patients:
  Complete Response (CR): Bone marrow: ≤ 5% myeloblasts with normal maturation. Peripheral blood: Hgb ≥ 11 g/dL Platelets ≥ 100 × 109/L Neutrophils ≥ 1.0 × 109/L, Blasts 0% Partial response (PR): All CR criteria if abnormal before treatment except: bone marrow blasts decreased by ≥ 50% over pretreatment but still > 5% Hematologic Improvement (HI): (responses must last at least 8 weeks) Erythroid response [HI-E; (if pretreatment Hgb < 11 g/dL)]; Hgb increase by ≥ 1.5 g/dL; Relevant reduction of units of red blood cell (RBC) transfusions by an absolute number of at least 4 RBC transfusions/8 weeks compared with the pretreatment transfusion number in the previous 8 weeks. Only RBC transfusions given for an Hgb of ≤ 9.0 g/dL pretreatment will count in the RBC transfusion response evaluation.
Number of AML patients with response | 171 Days (6 cycles of 28 days plus 3 day loading period)
  Complete Response (CR): Bone marrow: ≤ 5% myeloblasts with normal maturation of all cell lines, Absolute neutrophil count (ANC) >/= 1.0 X 109/L, platelet count >/= 100 X 109/L, no detectable Auer rods and no extramedulary leukemia.
  Complete Response (CR) with incomplete hematologic recovery (CRi): Responses as in CR but ANC < 1.0 X 109/L.
  Complete Response (CR) with incomplete platelets recovery (CRp): Responses as in CR but platelets < 100 X 109/L.
  Partial response (PR): All CR criteria if abnormal before treatment except: bone marrow blasts decreased by ≥ 50% over pretreatment but still > 5%.

SECONDARY OUTCOMES:
Incidence of adverse events | 171 Days (6 cycles of 28 days plus 3 day loading period)
  Incidence of adverse events of the combination defined by CTCAE 4.1 criteria. Toxicity will be any drug related Grade 3 or 4 toxicity.
Response duration | 171 Days (6 cycles of 28 days plus 3 day loading period)
  Response duration to the combination recorded from start of treatment to progression
Overall survival | Up to 1 year from end of treatment
  Overall survival measured from start of treatment to death or last follow up

CONTACTS AND LOCATIONS:
Overall Officials: Aziz Nazha, MD, Principal Investigator — Cleveland Clinic, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-05-24): https://cdn.clinicaltrials.gov/large-docs/73/NCT03397173/Prot_SAP_000.pdf
  • Informed Consent Form (2020-11-10): https://cdn.clinicaltrials.gov/large-docs/73/NCT03397173/ICF_001.pdf